CLINICAL TRIAL: NCT06943391
Title: CLINICAL STUDY OF BIOSTIMULATION WITH LOW-POWER DIODE LASER AFTER DENTAL EXTRACTIONS
Acronym: CSBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ID: 2934/2020
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Laser Therapy, Low-Level
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Intervention Model Description: Group I (Experimental): patients subjected to a tooth extraction and immediately given an intraoral PBM session with an EPIC X Biolase diode laser (BIOLASE, Inc. USA), with a voltage of 100-240 V, 1.5 A, a power of 0.5 W, and an application of an energy of 15J per cm², for 10-30 seconds at 1 mm of the tissue with an sterile surgical tip, based on the opti-mum biostimulation parameters by Cronshaw et al. . It was applied at three points in the area: buccal, palatal/lingual, and occlusal to stimulate the tissue. Group II (Sham): pa-tients undergoing tooth extraction and the application of inactive/simulated PBM imme-diately after using the same procedure
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Experimental): (Experimental): patients subjected to a tooth extraction and immediately given an intraoral PBM session with an EPIC X Biolase diode laser (BIOLASE, Inc. USA), . It was applied at three points in the area: buccal, pala-tal/lingual, and occlusal to stimulate the tissue
  Interventions: Device: laser
- Group Sham (Sham Comparator): patients undergoing tooth extraction and the application of inactive/simulated PBM im-mediately after using the same procedure
  Interventions: Device: laser

INTERVENTIONS:
Device: laser — patients subjected to a tooth extraction and immediately given an intraoral PBM session with an EPIC X Biolase diode laser (BIOLASE, Inc. USA), with a voltage of 100-240 V, 1.5 A, a power of 0.5 W, and an application of an energy of 15J per cm², for 10-30 seconds at 1 mm of the tissue with an sterile surgical tip. It was applied at three points in the area: buccal, pala-tal/lingual, and occlusal to stimulate the tissue.

SUMMARY:
the objective of the present work is to assess the efficacy of photobiomodulation (PBM) with respect to pain, inflammation, and healing after tooth extractions as compared with a sham treatment

ELIGIBILITY:
Inclusion criteria: adult patients who needed tooth extractions for any reason and who signed an informed consent form

Exclusion Criteria:patients who according to the ASA preoperative evaluation, did not meet the medical con-ditions for a surgical intervention. Immunocompromised patients. Patients with decom-pensated systemic diseases; undergoing chemotherapy treatment or taking immunosup-pressants. Pregnant women. Patients with severe mental disorders. Patients who had re-ceived head and neck radiotherapy

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-06-20 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (Self-Reported Visual Analog Scale - VAS, 0-10) | Self-reported Pain Scores Using 0m Visual Analog Scale 10 Pain Score.Total pain improvement over day 0 to day 7
  hange in self-reported pain scores from Day 0 to Day 7 using a 0-10 Visual Analog Scale (VAS), where 0 = no pain and 10 = worst imaginable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Lopez-Jornet Pia, Mur, Spain, Spain

REFERENCES:
- [Background] Ahrari F, Eshghpour M, Zare R, Ebrahimi S, Fallahrastegar A, Khaki H. Effectiveness of Low-Level Laser Irradiation in Reducing Pain and Accelerating Socket Healing After Undisturbed Tooth Extraction. J Lasers Med Sci. 2020 Summer;11(3):274-279. doi: 10.34172/jlms.2020.46. Epub 2020 Jun 21. PMID 32802287
- [Background] Camolesi GCV, Silva FFVE, Aulestia-Viera PV, Marichalar-Mendia X, Gandara-Vila P, Perez-Sayans M. IS THE PHOTOBIOMODULATION THERAPY EFFECTIVE IN CONTROLLING POST-SURGICAL SIDE EFFECTS AFTER THE EXTRACTION OF MANDIBULAR THIRD MOLARS? A SYSTEMATIC REVIEW AND META-ANALYSIS. J Evid Based Dent Pract. 2024 Jun;24(2):101983. doi: 10.1016/j.jebdp.2024.101983. Epub 2024 Feb 28. PMID 38821660